CLINICAL TRIAL: NCT03354117
Title: On Demand Contraception: Investigating Efficacy of Ulipristal Acetate Plus a COX-2 Inhibitor at Peak Fertility
Brief Title: On Demand Contraception: Ulipristal Acetate Plus a COX-2 Inhibitor at Peak Fertility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Erica Cahill, Clinical Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 43881
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Contraception
MeSH Terms: interventions — ulipristal acetate; Tablets; Meloxicam

STUDY DESIGN:
Intervention Model Description: Single, open-label trial of one-time dosing of ulipristal acetate and meloxicam at a peak fertility time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ulipristal 30mg plus Meloxicam 15mg (Experimental): Each study participant will complete one menstrual cycle without medication. Her second menstrual cycle, each study participant will receive ulipristal acetate plus meloxicam at peak fertility.
  Interventions: Drug: Ulipristal Acetate 30 MG Oral Tablet

INTERVENTIONS:
Drug: Ulipristal Acetate 30 MG Oral Tablet — Each study participant will receive one dose of the study medication (ulipristal acetate 30mg plus meloxicam 15mg) at peak fertility in the treatment cycle.
  Other Names: Meloxicam

SUMMARY:
This is an exploratory prospective study investigating if addition of a COX-2 inhibitor can increase efficacy of ulipristal in disrupting ovulation at peak fertility.

DETAILED DESCRIPTION:
This is an exploratory prospective study investigating if addition of a COX-2 inhibitor can increase efficacy of ulipristal in disrupting ovulation at peak fertility. We will compare the proportion of women with ovulatory disruption after taking the study medications with those women's own placebo cycles and also to previously established/published rates of ovulatory disruption of ulipristal alone.9 Given the established efficacy of ulipristal during the follicular time period as well as the theoretical mechanism of meloxicam to disrupt cumulus-oocyte expansion is a late step in ovulation, we hypothesize that this medication could emerge as the best candidate for an oral on-demand contraceptive option.

ELIGIBILITY:
Inclusion Criteria:

Women, aged 18-38

* English speaking
* Able to consent, literate
* Access to smart phone throughout study
* History of regular menses
* Documented baseline cycle with ovulation
* Not currently using or needing hormonal contraception
* Not currently using or needing regular NSAIDS
* Able to commit to frequency of study visits

Exclusion Criteria:

* Currently or recently (<2months) pregnant
* Currently or recent (<2months) breastfeeding
* Current or recent (<2months) use of hormonal medication
* Regular NSAID use
* Known cardiac risk factors (e.g. personal history of obesity, HTN, cardiac disease, diabetes)
* BMI > 30, as some studies have shown decreased efficacy of ulipristal in obese women37
* Allergy or previous unacceptable side effects with study medications

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is evaluating efficacy of these medications in prevention of ovulation.
Enrollment: 12 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
ovulatory disruption | 8 weeks from start of study, approximately
  (1) no follicle rupture or (2) follicle rupture that was (a) not preceded within 24-48 hours by an LH peak, (b) preceded by a blunted LH peak (<21IU/L), and/or (c) followed by a luteal phase progesterone peak of <3ng/mL

SECONDARY OUTCOMES:
luteal hormone levels | 8 weeks from start of study, approximately
  luteal hormone levels
progesterone hormone levels | 8 weeks from start of study, approximately
  progesterone hormone levels
maximum follicle diameter | 8 weeks from start of study, approximately
  maximum ovarian follicle diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cahill EP, Lerma K, Shaw KA, Blumenthal PD. Potential candidate for oral pericoital contraception: evaluating ulipristal acetate plus cyclo-oxygenase-2 inhibitor for ovulation disruption. BMJ Sex Reprod Health. 2022 Jul;48(3):217-221. doi: 10.1136/bmjsrh-2021-201446. Epub 2022 Apr 25. PMID 35470225